CLINICAL TRIAL: NCT05762185
Title: Interest of a Nursing Consultation in the Empowerment of the Patient With Rheumatoid Arthritis in the Management of His Subcutaneous Biotherapy
Acronym: PRECI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI2019_843_0045
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Biotherapies; Rheumatology; Rheumatoid Arthritis
Keywords: nurse consultation; biotherapies; Rheumatology; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nursing consultation (Experimental)
  Interventions: Device: nursing consultation

INTERVENTIONS:
Device: nursing consultation — nursing consultation

SUMMARY:
Biotherapy present specifics risks that patients must know and learn to manage. A national survey has been carried in this study to evaluate patients safety skills. (wording: " cross study of safety skills of 677 patients treat by biopharmaceuticals for an inflammatory rheumatism). This survey has allowed showcasing patients difficulties in managing their treatment, including for those under subcutaneous biotherapy. More than 60% patients interviewed doesn't know symptoms to bring them to consult and mainly postpone to their injection. The aim of this study is to prove that nursing consultation can allow the patient to become independent in treatment management and thus avoid occurrence of adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from rheumatoid arthritis followed by Rheumatology consultation of Amiens-Picardie University Hospital
* Patient treated by Subcutaneous Biotherapy for at least 6 months at the time of inclusion
* Major patient
* Patient having signed an informed consent

Exclusion Criteria:

* Minor patient
* Patient with cognitive impairment diagnosed by a physician
* Patient under tutorship or curatorship
* Patient deaf or hard of hearing
* Patient not fluent in the French language (at the decision of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Variation of BIOSECURE score between baseline and after nurse consultation | one day
  Biosecure questionnaire is assessing patient theoretical and practical understanding of biotherapy. Highest score is 100.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No